CLINICAL TRIAL: NCT04223791
Title: A Phase 3, Randomized, Active-Controlled, Double-Blind Clinical Study to Evaluate a Switch to Doravirine/Islatravir (DOR/ISL) Once-Daily in Participants With HIV-1 Virologically Suppressed on Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/FTC/TAF)
Brief Title: Switch to Doravirine/Islatravir (DOR/ISL) in Human Immunodeficiency Virus 1 (HIV-1) Participants Treated With Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/FTC/TAF) (MK-8591A-018)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8591A-018; MK-8591A-018 (Other: Merck); 205166 (Registry Identifier: JAPIC-CTI); 2019-000587-23 (EudraCT Number)
Record Dates: First submitted 2020-01-08; First posted 2020-01-10 (Actual); Results first posted 2022-08-22 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DOR/ISL (Experimental): A fixed dose combination (FDC) of 100 mg doravirine (DOR)/0.75 mg islatravir (ISL) for 144 weeks; and placebo to Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/FTC/TAF) for 96 weeks.
  Interventions: Drug: DOR/ISL; Drug: Placebo to BIC/FTC/TAF
- BIC/FTC/TAF (Active Comparator): 50 mg bictegravir (BIC), 200 mg emtricitabine (FTC), 25 mg tenofovir alafenamide (TAF) for 144 weeks, and placebo to FDC DOR/ISL for 96 weeks. Participants will be offered the option to receive open-label FDC DOR/ISL from Week 144 to Week 156.
  Interventions: Drug: DOR/ISL; Drug: BIC/FTC/TAF; Drug: Placebo to FDC DOR/ISL

INTERVENTIONS:
Drug: DOR/ISL — 100 mg DOR/ 0.75 ISL FDC tablet taken orally once daily
  Other Names: MK-8591A
Drug: BIC/FTC/TAF — 50 mg BIC, 200 mg FTC, and 25 mg TAF combined in a single tablet, taken orally once daily
  Arms: BIC/FTC/TAF
Drug: Placebo to BIC/FTC/TAF — Placebo to BIC/FTC/TAF in a single tablet taken orally, once daily
  Arms: DOR/ISL
Drug: Placebo to FDC DOR/ISL — Placebo to FDC DOR/ISL in a tablet taken orally, once daily
  Other Names: Placebo to MK-8591A
  Arms: BIC/FTC/TAF

SUMMARY:
This study will evaluate the safety and efficacy of a switch to MK-8591A (a fixed dose combination of doravirine and islatravir) in human immunodeficiency virus -1 (HIV-1)-infected participants virologically suppressed on a regimen of bictegravir/emtricitabine/tenofovir alafenamide (BIC/FTC/TAF). The primary hypothesis is that a switch to MK-8591A will be non-inferior to continued treatment with BIC/FTC/TAF as assessed by the proportion of participants with HIV-1 ribonucleic acid (RNA) ≥50 copies/mL at Week 48. Participants who benefit from their assigned intervention (as determined by investigator) will be able to continue treatment through a 24-week study extension.

ELIGIBILITY:
Inclusion Criteria:

* Is HIV-1 positive with plasma Human Immunodeficiency Virus 1 (HIV-1) RNA <50 copies/mL at screening.
* Has been receiving BIC/FTC/TAF therapy with documented viral suppression (HIV-1 RNA <50 copies/mL) for ≥3 months prior to signing informed consent and has no history of prior virologic treatment failure on any past or current regimen.
* Female is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies: Is not a woman of childbearing potential (WOCBP); is a WOCBP and using an acceptable contraceptive method, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle; a WOCBP must have a negative highly sensitive pregnancy test ([urine or serum] as required by local regulations) within 24 hours before the first dose of study intervention; if a urine test cannot be confirmed as negative (e.g. an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.

Exclusion Criteria:

* Has HIV-2 infection.
* Has an active diagnosis of hepatitis due to any cause, including active Hepatitis B Virus (HBV) co-infection.
* Has a history of malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or cutaneous Kaposi's sarcoma.
* Is taking or is anticipated to require systemic immunosuppressive therapy, immune modulators, or any prohibited therapies.
* Is currently participating in or has participated in a clinical study with an investigational compound or device from 45 days prior to Day 1 through the study treatment period.
* Has a documented or known virologic resistance to DOR.
* Female expects to conceive or donate eggs at any time during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2021-08-26 (Actual); Study Completion 2025-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (89):
- United States (28):
  - Pueblo Family Physicians ( Site 2717), Phoenix, Arizona
  - Pacific Oaks Medical Group ( Site 2765), Beverly Hills, California
  - Men's Health Foundation ( Site 2749), Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center ( Site 2775), Los Angeles, California
  - Eisenhower Medical Center ( Site 2744), Palm Springs, California
  - University of California, Davis, Division of ID Research ( Site 2702), Sacramento, California
  - Zuckerberg San Francisco General Hospital UCSF ( Site 2743), San Francisco, California
  - Whitman-Walker Clinic ( Site 2728), Washington D.C., District of Columbia
  - TheraFirst Medical Center ( Site 2742), Fort Lauderdale, Florida
  - Midway Immunology and Research ( Site 2759), Ft. Pierce, Florida
  - The Kinder Medical Group ( Site 2739), Miami, Florida
  - AHF South Beach ( Site 2780), Miami Beach, Florida
  - Orlando Immunology Center ( Site 2734), Orlando, Florida
  - Triple O Research Institute, P.A. ( Site 2755), West Palm Beach, Florida
  - Augusta University ( Site 2752), Augusta, Georgia
  - Infectious Disease Specialists Of Atlanta PC ( Site 2719), Decatur, Georgia
  - Mercer University ( Site 2738), Macon, Georgia
  - Chatham County Health Department ( Site 2731), Savannah, Georgia
  - Hennepin County Medical Center ( Site 2733), Minneapolis, Minnesota
  - Kansas City CARE Clinic ( Site 2718), Kansas City, Missouri
  - ID Care ( Site 2751), Hillsborough, New Jersey
  - Icahn School of Medicine at Mount Sinai ( Site 2700), New York, New York
  - Montefiore Einstein Center ( Site 2730), The Bronx, New York
  - North Texas ID Consultants, PA ( Site 2707), Dallas, Texas
  - The Crofoot Research Center, Inc. ( Site 2715), Houston, Texas
  - DCOL Center for Clinical Research ( Site 2769), Longview, Texas
  - Dr. Peter Shalit, MD ( Site 2770), Seattle, Washington
  - Multicare Health System ( Site 2713), Spokane, Washington
- Australia (7):
  - St Vincent's Hospital ( Site 3807), Darlinghurst, New South Wales
  - Taylor Square Private Clinic ( Site 3804), Darlinghurst, New South Wales
  - Holdsworth House Medical Practice ( Site 3800), Sydney, New South Wales
  - Holdsworth House Medical Practice - Brisbane ( Site 3810), Brisbane, Queensland
  - Royal Brisbane and Womens Hospital- Infectious Diseases Unit ( Site 3812), Herston, Queensland
  - The Alfred Hospital ( Site 3802), Melbourne, Victoria
  - Prahran Market Clinic (PMC) ( Site 3806), Melbourne, Victoria
- Austria (4):
  - LKH Graz West ( Site 3401), Graz, Styria
  - Medical University Vienna ( Site 3402), Vienna, Vienna
  - Sozialmedizinisches Zentrum Sued - Kaiser-Franz-Josef-Spital ( Site 3400), Vienna, Vienna
  - Social Medical Center - Otto Wagner Hospital ( Site 3404), Vienna, Vienna
- Canada (4):
  - Vancouver ID Research and Care Centre Society ( Site 2800), Vancouver, British Columbia
  - Hamilton Health Sciences ( Site 2803), Hamilton, Ontario
  - Clinique de Medecine Urbaine du Quartier Latin ( Site 2804), Montreal, Quebec
  - Clinique Medicale L Actuel ( Site 2814), Montreal, Quebec
- Helsinki University Hospital ( Site 3200), Helsinki, Uusimaa, Finland
- France (12):
  - Hopital Edouard Herriot ( Site 3126), Lyon, Ain
  - CHU de Nice Hopital Archet 1 ( Site 3103), Nice, Alpes-Maritimes
  - Hopital Europeen Marseille ( Site 3117), Marseille, Bouches-du-Rhone
  - Hopital Foch ( Site 3129), Suresnes, Hauts-de-Seine
  - CHU de Montpellier - Hopital Saint-Eloi ( Site 3121), Montpellier, Herault
  - CHU Hotel Dieu Nantes ( Site 3120), Nantes, Loire-Atlantique
  - Centre Hospitalier Regional du Orleans ( Site 3108), Orléans, Loiret
  - CHU de Nancy Hopital Brabois Adultes ( Site 3128), Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Centre Hospitalier de Tourcoing ( Site 3100), Tourcoing, Nord
  - Hopital Saint-Antoine ( Site 3113), Paris
  - Hopital Pitie Salpetriere ( Site 3111), Paris
  - Hopital Tenon ( Site 3118), Paris
- Germany (11):
  - MVZ Karlsplatz Dr.med.Hans Jaeger ( Site 3002), Munich, Bavaria
  - Klinikum der LMU München ( Site 3004), Munich, Bavaria
  - Klinikum rechts der Isar der Technischen Universitat ( Site 3005), Munich, Bavaria
  - Infektiologikum ( Site 3001), Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover ( Site 3012), Hanover, Lower Saxony
  - Universitaetsklinikum Bonn ( Site 3000), Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Essen ( Site 3007), Essen, North Rhine-Westphalia
  - ZIBP-Zentrum fur Infektiologie Berlin Prenzlauer Berg GmbH ( Site 3003), Berlin
  - EPIMED GmbH ( Site 3008), Berlin
  - ICH Study Center GmbH & Co.KG ( Site 3009), Hamburg
  - Universitaetsklinikum Hamburg- Eppendorf (UKE) ( Site 3010), Hamburg
- Italy (5):
  - Fondazione IRCCS Ca' Granda-Ospedale Maggiore Policlinico ( Site 3501), Milan, Lombardy
  - Universita' Vita Salute. Ospedale San Raffaele ( Site 3502), Milan
  - Azienda Ospedaliera San Paolo ( Site 3503), Milan
  - ASST Fatebenefratelli-Ospedale Sacco ( Site 3500), Milan
  - A.O.R.N. dei Colli - Ospedale Cotugno ( Site 3507), Napoli
- Japan (3):
  - National Hospital Organization Nagoya Medical Center ( Site 7203), Nagoya, Aichi-ken
  - National Hospital Organization Osaka National Hospital ( Site 7202), Osaka
  - Center Hospital of the National Center for Global Health and Medicine ( Site 7201), Tokyo
- Puerto Rico (4):
  - CAIMED Center - Ponce School of Medicine ( Site 2903), Ponce
  - Puerto Rico CONCRA ( Site 2904), Rio Piedras
  - Clinical Research Puerto Rico Inc ( Site 2900), San Juan
  - Hope Clinical Research, Inc. ( Site 2902), San Juan
- Spain (10):
  - Hospital Universitari Germans Trias i Pujol ( Site 3601), Badalona, Barcelona [Barcelona]
  - Hospital Universitari Vall d Hebron ( Site 3602), Barcelona, Barcelona [Barcelona]
  - Hospital Universitari de Bellvitge ( Site 3612), LHospitalet de Llobregat, Barcelona [Barcelona]
  - Hospital Clinic i Provincial ( Site 3600), Barcelona
  - Hospital General Universitario Gregorio Maranon ( Site 3603), Madrid
  - Hospital Universitario Infanta Leonor ( Site 3606), Madrid
  - Hospital Universitario Ramon y Cajal ( Site 3611), Madrid
  - Hospital 12 de Octubre de Madrid ( Site 3605), Madrid
  - Hospital Universitario La Paz ( Site 3604), Madrid
  - Hospital Universitario Virgen de la Victoria ( Site 3609), Málaga

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Mills AM, Rizzardini G, Ramgopal MN, Osiyemi OO, Bogner JR, Hagins DP, Paredes R, Reynes J, Rockstroh JK, Carr A, Su FH, Klopfer SO, Eves K, Plank RM, Correll T, Fox MC. Switch to fixed-dose doravirine (100 mg) with islatravir (0.75 mg) once daily in virologically suppressed adults with HIV-1 on bictegravir, emtricitabine, and tenofovir alafenamide: 48-week results of a phase 3, randomised, controlled, double-blind, non-inferiority trial. Lancet HIV. 2024 Jun;11(6):e357-e368. doi: 10.1016/S2352-3018(24)00030-4. Epub 2024 May 8. PMID 38734016
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DOR/ISL | BIC/FTC/TAF
Started | 322 | 321
Treated | 322 | 319
Completed | 0 | 0
Not Completed | 322 | 321
Not completed — Lost to Follow-up | 0 | 4
Not completed — Physician Decision | 5 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 10 | 12
Not completed — Pregnancy | 1 | 1
Not completed — Ongoing in Study | 305 | 302

BASELINE CHARACTERISTICS:
Groups:
- DOR/ISL: An FDC of 100 mg DOR/0.75 mg ISL for 144 weeks; and placebo to BIC/FTC/TAF for 96 weeks.
- BIC/FTC/TAF: 50 mg BIC, 200 mg FTC, 25 mg TAF for 144 weeks, and placebo to FDC DOR/ISL for 96 weeks. Participants will be offered the option to receive open-label FDC DOR/ISL from Week 144 to Week 156.
- Total: Total of all reporting groups
Arm/Group | DOR/ISL | BIC/FTC/TAF | Total
Number analyzed (Participants) | 322 | 321 | 643
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.6 (12.6) | 48.0 (11.8) | 47.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 78 | 183
  Male | 217 | 243 | 460
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 64 | 55 | 119
  Not Hispanic or Latino | 256 | 261 | 517
  Unknown or Not Reported | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 14 | 13 | 27
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 58 | 56 | 114
  White | 240 | 240 | 480
  More than one race | 5 | 7 | 12
  Unknown or Not Reported | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Participants With Human Immunodeficiency Virus 1 Ribonucleic Acid (HIV-1 RNA) ≥50 Copies/mL at Week 48
Description: The Abbott RealTime PCR assay with a reliable lower limit of quantification of 40 copies/mL was used to measure the HIV-1 RNA level in blood samples obtained at each visit. The percentage of participants with HIV-1 RNA ≥50 copies/mL at Week 48 is presented using the FDA Snapshot missing data approach.
Time Frame: Week 48
Population: All participants who received ≥1 dose of study intervention. Participants were included in the treatment group to which they were randomized.
Measure: Number; unit: Percentage of Participants
Arm/Group | DOR/ISL | BIC/FTC/TAF
Number analyzed (Participants) | 322 | 319
Percentage of Participants | 0.6 | 0.3
Statistical Analysis 1: Comparison: DOR/ISL vs BIC/FTC/TAF; Test type: Non-Inferiority — Non-inferiority is concluded if the upper bound of the 2-sided multiplicity-adjusted 95% CI for the difference in the percentage of participants with HIV-1 RNA ≥50 copies/mL (DOR/ISL-BIC/FTC/TAF) is less than 4 percentage points; p < .001, Unstratified Miettinen and Nurminen — p-value for the treatment differences in percent response were calculated using the unstratified Miettinen and Nurminen method; Estimated difference = 0.31, 95% CI 2-sided [-1.19 to 1.96] — Treatment difference for DOR/ISL group-BIC/FTC/TAF group

2. Primary Outcome: Percentage of Participants With One or More Adverse Events (AEs) up to Week 48
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who experienced an AE up to week 48 is presented.
Time Frame: Up to 48 weeks
Population: All randomized participants who received ≥1 dose of study intervention. Participants were included in the treatment group corresponding to the study intervention received.
Measure: Number; unit: Percentage of Participants
Arm/Group | DOR/ISL | BIC/FTC/TAF
Number analyzed (Participants) | 322 | 319
Percentage of Participants | 71.1 | 74.6
Statistical Analysis 1: Comparison: DOR/ISL vs BIC/FTC/TAF; Test type: Other — Difference between treatment groups; Difference in % (DOR/ISL- BIC/FTC/TAF) = -3.5, 95% CI 2-sided [-10.4 to 3.4] — Based on Miettinen and Nurminen method

3. Primary Outcome: Percentage of Participants Who Discontinued Study Intervention Due to an AE up to Week 48
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The percentage of participants who discontinued study intervention due to an AE up to week 48 is presented.
Time Frame: Up to 48 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | DOR/ISL | BIC/FTC/TAF
Number analyzed (Participants) | 322 | 319
Percentage of Participants | 2.5 | 2.5
Statistical Analysis 1: Comparison: DOR/ISL vs BIC/FTC/TAF; Test type: Other — Difference between treatment groups; Difference in % (DOR/ISL- BIC/FTC/TAF) = -0.02, 95% CI 2-sided [-2.7 to 2.6] — Based on Miettinen and Nurminen method

4. Secondary Outcome: Participants With HIV-1 RNA ≥50 Copies/mL at Week 96
Description: The Abbott RealTime PCR assay with a reliable lower limit of quantification of 40 copies/mL was used to measure the HIV-1 RNA level in blood samples obtained at each visit. The percentage of participants with HIV-1 RNA ≥50 copies/mL at Week 96 is presented.
Time Frame: Week 96
Reporting Status: Not Posted, anticipated posting 2026-02

5. Secondary Outcome: Participants With HIV-1 RNA ≥50 Copies/mL at Week 144
Description: The Abbott RealTime PCR assay with a reliable lower limit of quantification of 40 copies/mL was used to measure the HIV-1 RNA level in blood samples obtained at each visit. The percentage of participants with HIV-1 RNA ≥50 copies/mL at Week 144 is presented.
Time Frame: Week 144
Reporting Status: Not Posted, anticipated posting 2026-02

6. Secondary Outcome: Percentage of Participants With HIV-1 RNA <50 Copies/mL at Week 48
Description: The Abbott RealTime PCR assay with a reliable lower limit of quantification of 40 copies/mL was used to measure the HIV-1 RNA level in blood samples obtained at each visit. The percentage of participants with HIV-1 RNA <50 copies/mL at Week 48 is presented using the FDA snapshot missing data approach
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | DOR/ISL | BIC/FTC/TAF
Number analyzed (Participants) | 322 | 319
Percentage of Participants | 93.8 | 94.4

7. Secondary Outcome: Percentage of Participants With HIV-1 RNA <40 Copies/mL at Week 48
Description: The Abbott RealTime PCR assay with a reliable lower limit of quantification of 40 copies/mL was used to measure the HIV-1 RNA level in blood samples obtained at each visit. The percentage of participants with HIV-1 RNA <40 copies/mL at Week 48 is presented using the FDA snapshot missing data approach.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | DOR/ISL | BIC/FTC/TAF
Number analyzed (Participants) | 322 | 319
Percentage of Participants | 93.2 | 94.0

8. Secondary Outcome: Participants With HIV-1 RNA <40 or <50 Copies/mL at Week 96
Description: The Abbott RealTime PCR assay with a reliable lower limit of quantification of 40 copies/mL was used to measure the HIV-1 RNA level in blood samples obtained at each visit. The percentage of participants with HIV-1 RNA <40 or <50 copies/mL at Week 96 is presented.
Time Frame: Week 96
Reporting Status: Not Posted, anticipated posting 2026-02

9. Secondary Outcome: Participants With HIV-1 RNA <40 or <50 Copies/mL at Week 144
Description: The Abbott RealTime PCR assay with a reliable lower limit of quantification of 40 copies/mL was used to measure the HIV-1 RNA level in blood samples obtained at each visit. The percentage of participants with HIV-1 RNA <40 or <50 copies/mL at Week 144 is presented.
Time Frame: Week 144
Reporting Status: Not Posted, anticipated posting 2026-02

10. Secondary Outcome: Change From Baseline in Cluster of Differentiation-positive (CD4+) T-cell Count at Week 48
Description: Blood samples were used to measure CD4+ T-cell count. Baseline measurement of CD4+ T-cell count is defined as the day 1 value for each participant. Change from baseline in CD4+ T-cell count at week 48 using the data as observed (DAO) approach is presented. A negative value indicates a mean decrease in CD4+ T-cell count from baseline and a positive value indicates a mean increase in CD4+ T-cell count from baseline.
Time Frame: Baseline and Week 48
Population: All participants who received ≥1 dose of study intervention and who had baseline data for CD4+ T-cell count. Participants were included in the treatment group to which they were randomized.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | DOR/ISL | BIC/FTC/TAF
Number analyzed (Participants) | 301 | 298
cells/mm^3 | -19.66 [-39.78 to 0.45] | 40.51 [20.66 to 60.36]

11. Secondary Outcome: Change From Baseline in CD4+ T-cell Count at Week 96
Description: Blood samples were used to measure CD4+ T-cell count. Baseline measurement of CD4+ T-cell count is defined as the day 1 value for each participant. Change from baseline in CD4+ T-cell count at week 96 using the data as observed (DAO) approach is presented. A negative value indicates a mean decrease in CD4+ T-cell count from baseline and a positive value indicates a mean increase in CD4+ T-cell count from baseline.
Time Frame: Baseline and Week 96
Reporting Status: Not Posted, anticipated posting 2026-02

12. Secondary Outcome: Change From Baseline in CD4+ T-cell Count at Week 144
Description: Blood samples were used to measure CD4+ T-cell count. Baseline measurement of CD4+ T-cell count is defined as the day 1 value for each participant. Change from baseline in CD4+ T-cell count at week 144 using the data as observed (DAO) approach is presented. A negative value indicates a mean decrease in CD4+ T-cell count from baseline and a positive value indicates a mean increase in CD4+ T-cell count from baseline.
Time Frame: Baseline and Week 144
Reporting Status: Not Posted, anticipated posting 2026-02

13. Secondary Outcome: Participants With Viral Drug Resistance-associated Substitutions at Week 48
Description: Viral drug resistance is defined as participants with confirmed HIV-1 RNA ≥400 copies/mL having genotypic or phenotypic evidence of resistance to the study drug administered. The number of participants who demonstrate drug resistance is presented.
Time Frame: Week 48
Population: Participants who met the definition of confirmed virologic rebound (two consecutive [2 to 4 weeks apart] occurrences of HIV-1 RNA ≥200 copies/mL) at any time during the study or who discontinued study intervention for another reason and have HIV-1 RNA ≥200 copies/mL at the time of discontinuation. Participants for whom available genotypic or phenotypic data showed evidence of resistance, irrespective of viral load, were also included.
Measure: Count of Participants; unit: Participants
Arm/Group | DOR/ISL | BIC/FTC/TAF
Number analyzed (Participants) | 1 | 0
Participants | 0 |

14. Secondary Outcome: Participants With Evidence of Viral Drug Resistance-associated Substitutions at Week 96
Description: Viral drug resistance is defined as participants with confirmed HIV-1 RNA ≥400 copies/mL and/or genotypic or phenotypic analysis of data showing evidence of resistance to the study drug administered. The number of participants who demonstrate drug resistance is presented.
Time Frame: Week 96
Reporting Status: Not Posted, anticipated posting 2026-02

15. Secondary Outcome: Participants With Evidence of Viral Drug Resistance-associated Substitutions at Week 144
Description: as for outcome 14
Time Frame: Week 144
Reporting Status: Not Posted, anticipated posting 2026-02

16. Secondary Outcome: Change From Baseline in Body Weight at Week 48
Description: Body weight was measured and recorded at baseline and week 48. Participants removed their shoes and wore a single layer of clothing at each measurement. The mean change from baseline in body weight at week 48 is presented.
Time Frame: Baseline and Week 48
Population: Participants who received ≥1 dose of study intervention and were included in the treatment group corresponding to the study intervention received. The analysis population included participants with baseline and at least one postbaseline test result in the specified analysis window.
Measure: Mean (Standard Deviation); unit: kilogram (kg)
Arm/Group | DOR/ISL | BIC/FTC/TAF
Number analyzed (Participants) | 306 | 302
kilogram (kg) | 0.23 (4.19) | 0.55 (4.40)
Statistical Analysis 1: Comparison: DOR/ISL vs BIC/FTC/TAF; Test type: Superiority; p = 0.392, ANCOVA; Model included terms for baseline weight, sex, race, and treatment; Treatment Difference = -0.30, 95% CI 2-sided [-0.99 to 0.39] — Treatment difference for DOR/ISL group-BIC/FTC/TAF group

17. Secondary Outcome: Change From Baseline in Body Weight at Week 96
Description: Body weight was measured and recorded at baseline and week 96. Participants removed their shoes and wore a single layer of clothing at each measurement.
Time Frame: Baseline and Week 96
Reporting Status: Not Posted, anticipated posting 2026-02

18. Secondary Outcome: Change From Baseline in Body Weight at Week 144
Description: Body weight was measured and recorded at baseline and week 144. Participants removed their shoes and wore a single layer of clothing at each measurement.
Time Frame: Baseline and Week 144
Reporting Status: Not Posted, anticipated posting 2026-02

19. Secondary Outcome: Percentage of Participants With One or More AEs up to Week 144
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Time Frame: Up to Week 144
Reporting Status: Not Posted, anticipated posting 2026-02

20. Secondary Outcome: Percentage of Participants Who Discontinued Study Intervention Due to an AE up to Week 144
Description: as for outcome 19
Time Frame: Up to Week 144
Reporting Status: Not Posted, anticipated posting 2026-02

ADVERSE EVENTS:
Time Frame: Up to 48 weeks
Description: All-cause mortality population includes all randomized participants in their planned treatment groups. Adverse event population includes all randomized participants who received ≥1 dose of study intervention and were included in the treatment group corresponding to the study intervention received.
Arm/Group | DOR/ISL | BIC/FTC/TAF
All-Cause Mortality (participants affected / at risk) | 1/322 | 0/321
Serious Adverse Events (participants affected / at risk) | 13/322 | 15/319
Other Adverse Events (participants affected / at risk) | 71/322 | 80/319
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOR/ISL (N=322) | BIC/FTC/TAF (N=319)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Splenic artery aneurysm (Gastrointestinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis escherichia (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Neurosyphilis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brachial plexopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DOR/ISL (N=322) | BIC/FTC/TAF (N=319)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 20 (21)
COVID-19 (Infections and infestations) | 18 (18) | 18 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 (22) | 19 (21)
Back pain (Musculoskeletal and connective tissue disorders) | 13 (14) | 17 (17)
Headache (Nervous system disorders) | 25 (42) | 23 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT04223791/Prot_SAP_000.pdf